CLINICAL TRIAL: NCT02530697
Title: The Association of Miltefosine and Pentoxifylline to Treat Mucosal and Cutaneous Leishmaniasis: An Open-label, Randomized Clinical Trial in Brazil
Brief Title: The Association of Miltefosine and Pentoxifylline to Treat Mucosal and Cutaneous Leishmaniasis: A Clinical Trial in Brazil
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, SOFIA SALES MARTINS, MD, PhD, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40068714.1.0000.5558
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Leishmaniasis
Keywords: Leishmaniasis; Mucocutaneous; Miltefosine; Pentoxifylline
MeSH Terms: conditions — Leishmaniasis | interventions — Meglumine Antimoniate; miltefosine; Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - Mucosal Antimoniate and Pentoxifylline (Active Comparator): 20mgSb+5/kg/day meglumine antimoniate intravenous for 28 days. Pentoxifylline 400mg 3x/daily for 28 days.
  Interventions: Drug: Meglumine antimoniate; Drug: Pentoxifylline
- Group 2 - Mucosal Miltefosine and Pentoxifylline (Experimental): Oral Miltefosine 2,5mg/kg/day up to 50mg 2x/daily. Oral Pentoxifylline 400mg 3x/daily for 28 days.
  Interventions: Drug: Miltefosine; Drug: Pentoxifylline
- Group 3 - Cutaneous Antimoniate and Pentoxifylline (Experimental): 20mgSb+5/kg/day meglumine antimoniate intravenous for 20 days Oral Pentoxifylline 400mg 3x/daily for 20 days.
  Interventions: Drug: Meglumine antimoniate; Drug: Pentoxifylline
- Group 4 - Cutaneous Miltefosine and Pentoxifylline (Experimental): Oral Miltefosine 2,5mg/kg/day up to 50mg 2x/daily Oral Pentoxifylline 400mg 3x/daily for 20 days.
  Interventions: Drug: Miltefosine; Drug: Pentoxifylline

INTERVENTIONS:
Drug: Meglumine antimoniate — 20mgSb+5/kg/day meglumine antimoniate intravenous for 28 days.
  Arms: Group 1 - Mucosal Antimoniate and Pentoxifylline; Group 3 - Cutaneous Antimoniate and Pentoxifylline
Drug: Miltefosine — Miltefosine 2,5mg/kg/day up to 50mg 2x/daily.
  Other Names: Miltefosnine
  Arms: Group 2 - Mucosal Miltefosine and Pentoxifylline; Group 4 - Cutaneous Miltefosine and Pentoxifylline
Drug: Pentoxifylline — Pentoxifylline 20mg/kg/day up to 400mg 3x/daily for 28 days.

SUMMARY:
Mucocutaneous leishmaniasis is endemic in the central region of Brazil and other countries worldwide. The standard treatment with meglumine antimoniate has a high rate of important adverse effects. This interventional study consists in a randomized clinical trial to access efficacy and safety of the association of miltefosine and pentoxifylline compared to meglumine antimoniate and pentoxifyline.

ELIGIBILITY:
Inclusion Criteria:

* Mucosal and/or cutaneous leishmaniasis, not treated or at least 6 months without any treatment to leishmaniasis;
* For patients with cutaneous lesions: duration of disease longer then a 1 month and shorter then 4 yeas; 1 to 3 lesions; larger lesions from 10mm to 50mm;
* Ages between 18 and 80 years old;
* Fertile female patients should use at least two contraceptive methods (hormonal and barrier);
* Agree to participate in the study and sign the informed consent term.

Exclusion Criteria:

* Use of any leishmanicidal drugs six months prior;
* Clinical or laboratorial evidences of electrocardiographic disorders;
* Renal, hepatic, cardiac diseases, uncontrolled diabetes or AIDS;
* Hypersensitivity to meglucamine antimoniate;
* Pregnancy or lactation;
* Fertile females that do not agree to use contraceptive methods;
* Patients that do not agree to the informed consent term.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Cure | 90 days
  Complete healing of previous lesions until the 90th day after the begin of the treatment
Failure | 90 days
  Lesions fail to heal until the 90th day after the begin of the treatment
Relapse | 90 days
  Lesions that reappear on the scar of a previously healed lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário de Brasília, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No